CLINICAL TRIAL: NCT06498232
Title: Effects of Structured Active Video Game-Based Exercise Training and Stabilization Training on Postural Control and Balance After Scoliosis Surgery in Adolescents
Brief Title: Active Video Game-Based Exercise Training and Stability Training After AIS Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AkyurekE1
Record Dates: First submitted 2024-06-27; First posted 2024-07-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Idiopathic Scoliosis; Spinal Fusion
Keywords: scoliosis; postural control; active video-based exercises; stabilization training; scoliosis surgery; post-op rehabilitation; balance
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I- Active Video Based Group (Experimental): Participants will play progressive, configured games with Nintendo Wii, supervised by a physiotherapist, 2 days a week for 12 weeks, for a total of 24 sessions. The game schedule will be divided into 4 phases: 1-3, 4-6, 7-9, and 10-12 weeks. Sessions will last 40 minutes in total, including 5 minutes of warm-up, 30 minutes of balance and sports games, and 5 minutes of cool-down.
  Interventions: Other: Active Video Based Exercises
- Group II- Exercise Group (Experimental): Participants will be included in a total of 24 sessions of progressive, configured exercise program, supervised by a physiotherapist, 2 days a week for 12 weeks. The exercise program will be divided into 4 phases: 1-3, 4-6, 7-9, and 10-12 weeks. Sessions will last 40 minutes in total, including 5 minutes of warm-up, 30 minutes of stabilization, strengthening, and balance exercises, and 5 minutes of cool-down.
  Interventions: Other: Stabilization and Strengthening Exercises
- Group III- Control Group (Other): Participants in the control group will be placed on a waiting list for 12 weeks. Participants in the control group will be given a 30-minute spine protection principles training and the things to pay attention to will be explained. Participants will not receive any exercise intervention for 12 weeks and will be able to continue their routine physical activities.
  Interventions: Other: Waiting List-Spine protection principles training

INTERVENTIONS:
Other: Active Video Based Exercises — Warm-up and cool-down will consist of aerobic games (Step, Hula Hoop, Rhythm Parade Dance, Run) available in Nintendo Wii. Balance games will consist of Penguin Slide, Soccer Heading, Table Tilt, Balance Bubble, Ski Slalom, Ski Jump, Tilt City, and Snowboard Slalom. Among the sports games, Bowling, Boxing, Tennis, and Baseball will be included in the program. In all games, progress will be made by increasing the difficulty levels, and in balance games, the game will be made more difficult with an additional balance board and bosu.
  Arms: Group I- Active Video Based Group
Other: Stabilization and Strengthening Exercises — Warm-up exercises will consist of active dynamic warm-up exercises. Stabilization and strengthening exercises; extremity movements will begin with teaching respiratory control in supine, prone, sitting, crawling, squat, and standing positions, and will be made more difficult with the addition of exercise tires and exercise balls. Balance exercises will start from static positions and move on to dynamic positions with the inclusion of different surfaces. In the cooling exercises, in addition to breathing exercises, stretching exercises will be performed for the trunk, upper and lower extremities.
  Arms: Group II- Exercise Group
Other: Waiting List-Spine protection principles training — Participants will be placed on a waiting list. Following the initial evaluations, participants will be informed that they will be included in an exercise program at the end of 6 months. During this process, participants in the control group will be called by phone at the 6th, 12th, and 18th weeks to question their status and to remind them that they will start the exercise program after a while. It will be evaluated at the end of 6 months, and the end of the study, exercise training approaches in the intervention group will be applied to participants who wish to do so, with the same protocol and duration.
  Arms: Group III- Control Group

SUMMARY:
The purpose of this clinical trial is to investigate the effects of "Active Video-Based Exercises (AVTE) on postural control and balance in comparison with stabilization exercises is (AIS) after Posterior Spinal Fusion (PSF) surgery. Fifty-one patients with AIS after PSF surgery will be randomly divided into groups as Group I-AVTE Group, Group II-Exercise Group, Group III-Control Group, and a 12-week program will be applied. Evaluations will be performed at baseline, 12 and 24 weeks. The primary evaluations will be postural stability and balance; secondary evaluations will be pain, trunk muscle strength, mobility, endurance, core stabilization, function, quality of life, and satisfaction.

DETAILED DESCRIPTION:
Posterior Spinal Fusion (PSF) is considered the gold standard in the surgical treatment of Adolescent Idiopathic Scoliosis (AIS) as it provides successful results in terms of deformity correction. However, it has been emphasized in many studies that postoperative rehabilitation should be planned to reduce pain and movement limitations of individuals after surgery and to increase their activity and participation levels. It is stated that postoperative rehabilitation programs should especially include stabilization, proprioception, and postural balance training. Postoperative rehabilitation after spinal surgery can consist of "stabilization exercises" or can be done with "Active Video-Based Exercises (AVTE)". However, no study was found in the literature investigating the effects of these two methods on postural control and balance in AIS patients who underwent PSF surgery. The primary aim of the study is to investigate the effects of AVTE on postural control and balance in comparison with stabilization exercises in patients with AIS after PSF surgery. The secondary purpose of these exercise trainings is; to comparatively examine its effects on pain, trunk muscle strength, mobility, endurance, core stabilization, function, quality of life, and satisfaction. It is thought that this study may be an effective, innovative, technology-based approach that will contribute to the improvement of postoperative postural control and balance in AIS patients.

Cases that meet the inclusion criteria of the study will be divided into 3 groups by randomization. These groups are Group 1: Video-Based Exercise Group, Group 2: Stabilization Exercise Group, Group 3: Control Group.

The participants included in the study will be evaluated as described below. Primary evaluation parameters; There will be postural stability and static and dynamic balance. Secondary evaluation parameters will be pain, trunk mobility, muscle strength, endurance, core stabilization, functional level, physical activity level, quality of life, and satisfaction. All evaluations will be performed by an investigator blinded to the intervention method.

Participants in the experimental group will receive a total of 24 sessions of Video-Based Exercise or Stabilization Exercise treatment, 2 days a week, for 12 weeks, under the supervision of a physiotherapist, while participants in the control group will be placed on a waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Adolescent Idiopathic Scoliosis by an orthopedic specialist
* Being between the ages of 10 and 18
* The Cobb angle determined on the anteroposterior radiograph must be over 45 degrees before surgery.
* Having had posterior spinal fusion surgery
* Between 8th week and 6 months postoperatively
* Ability to understand and follow instructions
* Volunteering to participate in the study

Exclusion Criteria:

* Complications that prevent rehabilitation after surgery (such as postoperative cerebrospinal fluid leak, paraparesis, hemiparesis)
* Neuromuscular, rheumatic disease or vestibular problems that may affect balance, vision-related diseases
* Orthopedic problems that may prevent participation in the exercise program
* Serious lung complications associated with surgery
* Any other exercise or physical activity that may affect trunk muscle strength or balance
* Patients who cannot understand and follow instructions

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Postural Stability Test | 12 weeks, 6 months
  The postural stability of the participants will be evaluated with the "Postural Stability Test" on a static surface via the postural stability assessment system.
Stability Limits Test | 12 weeks, 6 months
  The postural stability of the participants will be evaluated with the "Stability Limits Test" on a static surface via the postural stability assessment system.
Sensory Integration Test | 12 weeks, 6 months
  The static and dynamic balance of the participants will be evaluated with the "Sensory Integration Test" via the postural stability assessment system.
One-Legged Posture Test | 12 weeks, 6 months
  The static and dynamic balance of the participants will be evaluated with the "One-Legged Posture Test" via the postural stability assessment system.

SECONDARY OUTCOMES:
Spine Pain | 12 weeks, 6 months
  Numerical Pain Scale, which is frequently preferred by clinicians in determining and monitoring pain severity, will be used in pain assessment because it is easily applicable, can be done in a short time, can be repeated and the test is easy to understand. In this scale, patients will be asked to score the severity of their pain between 0 and 10, where 0 means "no pain" and 10 means "unbearable pain."
The forward bending test | 12 weeks, 6 months
  The forward bending test will be used to evaluate trunk flexibility in the sagittal plane. The patient is asked to sit tall on a hard surface with both knees extended, feet 15 cm apart from each other, leaning on a 25 cm long step, and reach the feet with his hands while his elbows are extended without flexing his knees. The distance between the third finger and the foot will be measured with a ruler and recorded as "cm".
The side bending test | 12 weeks, 6 months
  The side bending test will be used to evaluate trunk flexibility in the frontal plane. During the test, the patient will be asked to lean to the right and left side respectively, without leaving his back to the wall. The distance between the third finger and the ground will be measured with the help of a 50 cm long rigid ruler and recorded in "cm".
  In all evaluation sessions, each measurement will be repeated three times by the same physiotherapist, and the average of the measurements.
Trunk Isometric Muscle Strength | 12 weeks, 6 months
  Evaluation of trunk flexion, extension, and right-left lateral flexion isometric muscle strength will be performed with a manual muscle testing device, which is an objective, valid, and reliable method. Trunk flexion evaluation will be performed in the 30-degree supine position, trunk extension in the prone position, and lateral flexion in the sitting position.
Lateral Bridge Test | 12 weeks, 6 months
  One of the three trunk muscle endurance tests created by McGill, the lateral bridge test will be evaluated. Before the test, the required test position will be explained to the participant and he/she will be asked to try the appropriate position.
Trunk Extension Test | 12 weeks, 6 months
  One of the three trunk muscle endurance tests created by McGill, the trunk extension test will be evaluated. Before the test, the required test position will be explained to the participant and he/she will be asked to try the appropriate position.
Trunk Flexion Test | 12 weeks, 6 months
  One of the three trunk muscle endurance tests created by McGill, consisting of the trunk flexion test, will be evaluated. Before the test, the required test position will be explained to the participant and he/she will be asked to try the appropriate position.
Core Stabilization | 12 weeks, 6 months
  Core stabilization evaluation will be performed in supine and prone positions with the Stabilizer Pressure Feedback Unit. The "Shermann core stabilization test," which is valid and reliable in the supine position, will be used. This test consists of 5 increasingly difficult levels. The measurement will be repeated 3 times with 30-second rest periods, and the maximum value will be recorded.
Sock Test | 12 weeks, 6 months
  Valid and reliable sock test, will be used to evaluate the functional level of the cases.
  In the sock test, the patient will be asked to sit in a high place so that his feet do not touch the ground, and to lift one leg and put on the socks with both hands without his feet touching the chair. After testing each leg once, the patient will be given a score between 0-3. Lower values in the scoring will represent better performance.
Pick-up Test | 12 weeks, 6 months
  Valid and reliable pick-up test will be used to evaluate the functional level of the cases.
  In the picking test, the patient will be asked to pick up a piece of paper from the floor and the patient's performance will be evaluated using a 4-point ordinal scale. Lower values in the scoring will represent better performance.
Pebble Test | 12 weeks, 6 months
  Valid and reliable pebble test will be used to evaluate the functional level of the cases.
  In the pebble test, the participant will be asked to lift a 5 kg weight from the ground to the table (76 cm) and bring it back to the ground, and the number of lifts will be recorded.
Child Physical Activity Questionnaire (8-14 years old) | 12 weeks, 6 months
  The physical activity levels of the participants will be evaluated with the Child Physical Activity Questionnaire (8-14 years old), which provides valuable data and is valid and reliable in evaluating physical activity in healthy adolescents. Participants' high scores in the survey evaluation indicate that their physical activity levels have increased.
Adolescent Physical Activity Questionnaire (14-20 years old) | 12 weeks, 6 months
  The physical activity levels of the participants will be evaluated with the Adolescent Physical Activity Questionnaire (14-20 years old) which provides valuable data and is valid and reliable in evaluating physical activity in healthy adolescents. Participants' high scores in the survey evaluation indicate that their physical activity levels have increased.
Pedometer | 12 weeks, 6 months
  The physical activity levels of the participants will be evaluated with the pedometer, which provides objective data and is valid and reliable in evaluating physical activity in healthy adolescents. Participants will be instructed to wear the pedometer on their right or left hip side (non-dominant side) over their clothing or belt. The number of steps taken by participants during a week will be recorded. Participants' increase in the number of steps on the pedometer indicate that their physical activity levels have increased.
Scoliosis-Specific Quality of Life | 12 weeks, 6 months
  Scoliosis Research Society Questionnaire -30 (SRS-30) is a simple and practical quality of life questionnaire that is most frequently used to evaluate the quality of life in scoliosis patients and has been translated into our language and has validity and reliability, created specifically for individuals with scoliosis. Each question is scored from 1 (worst) to 5 (best) in the survey, which evaluates five domains: function, pain, self-image, mental health (five questions each), and treatment satisfaction (two questions).
Treatment Satisfaction | 12 weeks, 6 months
  Participants' satisfaction with the treatment will be evaluated with the Global Rating of Change (GRC). GRC is used quite frequently, especially in the field of the musculoskeletal system. This scale is designed to determine the extent of improvement or deterioration of the patient over time. It also indicates the effect of an intervention or the clinical course of a condition. In the GRC scale, the patient is asked to indicate the difference between their current health status and their health status before a specific point in time. The questions asked, the number of points on the scale, and the labels assigned to the scale points may vary. A 7-point scale (-3: much worse, -2: worse, -1: slightly worse, 0: the same, 1: slightly better, 2: quite better, 3: much better) will be used in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa; Turgut Akgül, Prof., Study Chair — Istanbul University; Elçin Akyurek, Msc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)